CLINICAL TRIAL: NCT03621176
Title: Effects of Home-based Exercise in Advanced Chronic Kidney Disease and End-stage Renal Disease
Brief Title: Home-based Exercise in Chronic Kidney Disease
Acronym: HBCKD-BCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Consorci Sanitari de Terrassa. Hospital de Terrassa (Unknown)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBCKD
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Disease; End-stage Renal Disease
Keywords: Exercise; Health-related quality of life; Physical function; Hemodialysis; Peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will undertake the exercise intervention. We will compare effects of the intervention between different cohorts included (advanced chronic kidney disease, end-stage renal disease hemodialysis o peritoneal dialysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based exercise (Experimental): Home-based intervention in the advanced chronic kidney disease group, hemodialysis or peritoneal dialysis group
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Home-based exercise — A booklet with detailed information will be provided, and the exercises will be previously reviewed with every patient by the researcher. Participants will be encouraged to perform at least 3 sessions per week and monitor their heart rate. They will be instructed that the exercises should be perceived as 'somewhat hard' from a rate of perceived exertion. Adaptations to increase the intensity of the exercises will be provided so that participants can progress in exercise intensity

SUMMARY:
A home-based exercise program will be implemented in three different groups of participants: advanced chronic kidney disease, end-stage renal disease in substitutive treatment hemodialysis or peritoneal dialysis. Participants will be evaluated before the program, after 3 months and after 6 months from the starting of the program. During the first 3 months the researcher will phone them weekly to reinforce the exercise habit, and during the last three months, there will be no reinforcement. Assessment will include strength, functional capacity, health-related quality of life and depressive symptoms.

DETAILED DESCRIPTION:
Three groups of participants (advanced chronic disease not yet in substitutive treatment, end-stage renal disease patients in hemodialysis and end-stage renal disease patients in peritoneal dialysis) will enter the study. The intervention will consist of a home-based exercise program. They will be provided with a booklet and the researcher will explain personally each of the exercises to the participants. Progression will be encouraged so that the participants should find the sessions 'somewhat hard' according to the rate of perceived exertion. Reinforcement will be high during the first 3 months (weekly phone calls, visits to the nephrology department) and none during the last 3 months. Assessment will be undertaken at three-time points: baseline, after 3 months of high reinforcement and after 3 more months of no reinforcement at all.

Assessment will include strength, functional capacity, health-related quality of life, cognitive state and depressive symptoms.

The aim of the study is to assess the effectiveness of home-based exercise to improve strength, physical function, health-related quality of life, cognitive state and depressive symptoms in advanced chronic kidney disease and end-stage renal disease (hemodialysis and peritoneal dialysis). We also aim at describing all these variables in the three different groups of patients. Adherence and satisfaction with the exercise program will be recorded at the end of the study.

Additionally, interobserver reliability will be calculated, so as reliability intraobserver in different measurement conditions (dialysis vs non-dialysis days).

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months in hemodialysis treatment
* Clinically stable

Exclusion Criteria:

* Recent cardiac events (less than 3 months)
* Unable to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline sit to stand 10 test at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Sit to stand to sit test 10, time to perform 10 repetitions

SECONDARY OUTCOMES:
Change from baseline Six-minute walking test at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Distance covered in 6 minutes
Change from baseline STS-60 at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Sit to stand to sit test 60, number of repetitions performed during 60 seconds
Change from baseline OLHR at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  One leg heel rise test, number of repetitions of heel rise to measure triceps strength
Change from baseline Handgrip strength (dynamometry) at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Handgrip strength measured through a dynamometer
Change from baseline SPPB at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Short physical performance battery, a combination of walking speed, STS-5 and balance
Change from baseline OLST at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  One-leg stand test, time to keep the balance in one leg
Change from baseline TUG at 12 and 24 weeks | Baseline,1 week, non-dialysis day baseline,12 weeks, 24 weeks
  Timed up and go test, time to stand up from a chair, walk 3m, turn around and sit back again
Change from baseline Albumin at 12 and 24 weeks | Baseline,12 weeks, 24 weeks
  Serum albumin in blood for dialysis patients
Change from baseline Health-related quality of life measured through the Euro quality of life questionnaire, 5 dimensions, at 12 and 24 weeks | Baseline,12 weeks, 24 weeks
  Euroquol 5D questionnaire, scale 0 (worst health) to 100 (best health). 5 Dimensions include mobility, personal care, activities of daily living, pain, and anxiety/depression
Change from baseline Beck depression inventory at 12 and 24 weeks | Baseline,12 weeks, 24 weeks
  Questionnaire to measure depressive symptoms. Range from 0 (normal) to 63 (worst depression)
Change from baseline Human activity profile at 12 and 24 weeks Human activity profile | Baseline,12 weeks, 24 weeks
  Questionnaire to measure physical activity. Higher score represents higher activity. Measures of average and maximal activity scores are reported. Average activity scores bellow 53 are considered impaired; between 53 and 74 are considered moderately active and above 74 are considered active.
Change from baseline Physical Activity Scale for the elderly at 12 and 24 weeks | Baseline,12 weeks, 24 weeks
  Questionnaire to measure physical activity. Higher scores represent higher activity.
Adherence | 12 weeks, 24 weeks
  Sessions performed/offered x 100

CONTACTS AND LOCATIONS:
Overall Officials: Vicent Esteve-Simó, PhD, Study Chair — Hospital de Terrassa
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteve Simo V, Junque Jimenez A, Moreno Guzman F, Carneiro Oliveira J, Fulquet Nicolas M, Pou Potau M, Saurina Sole A, Duarte Gallego V, Tapia Gonzalez I, Ramirez de Arellano M. Benefits of a low intensity exercise programme during haemodialysis sessions in elderly patients. Nefrologia. 2015;35(4):385-94. doi: 10.1016/j.nefro.2015.03.006. Epub 2015 Jul 21. English, Spanish. PMID 26306966
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637